CLINICAL TRIAL: NCT01714388
Title: Vagotonic Effect of Remifentanil in Reference to Sympathetic or Parasympathetic Predominance of Autonomic Nervous System.
Brief Title: Vagotonic Effect of Remifentanil and Autonomic Nervous System Activity.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Magdalena Wujtewicz, assistant professor, Medical University of Gdansk
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GUMed-Ow-004
Record Dates: First submitted 2012-10-23; First posted 2012-10-25 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Autonomic Nervous System Activity
Keywords: remifentanil; heart rate; autonomic nervous system; heart rate variability; autonomic nervous activity; vagotonic effect; single dose
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remifentanil, Vagotonic response (Experimental): 1 microgram/kg remifentanil given iv over at least 30 sec. at the beginning of induction of general anaesthesia
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — 1mcg/kg iv dose, followed by 5 minutes ECG recording
  Other Names: Ultiva

SUMMARY:
Remifentanil (RMFNT) is a very short active opioid, used for analgesia during general anaesthesia and for analgesic and sedative effect in intensive care units (ICU) patients. Registration for anesthesia includes bolus dose and continuous infusion, in ICU only infusion regimen is allowed. Pharmacokinetic/pharmacodynamic parameters of RMFNT results in rapid onset and offset of clinical effect, which makes this drug almost ideal in many situations. Unfortunately, its vagomimetic influence on cardiac activity may result in decrease of heart rate. It may be hypothesized that patients with parasympathetic predominance may be prone to more intense parasympathomimetic effect of this opioid. An optimal method for assessment of autonomic nervous system activity and assessment of influence of RMFNT on that activity is Heart Rate Variability (HRV) analysis. Parasympathetic predominance is expressed as high frequency (HF) power and HF/(LF+HF) (LF-low frequency) ratio in frequency domain and Root Mean Square of the Successive Difference (RMSSD), the number of pairs of successive NNs that differ by more than 50 ms (NN50), the proportion of NN50 divided by total number of NNs (pNN50) in time domain. The aim of this study is to verify the hypothesis that patients with predominance of parasympathetic activity are more subject to vagomimetic effect of RMFNT. HRV based on 5 minutes electrocardiogram (ECG) recorded before and after bolus dose of RMFNT will be analyzed. The occurrence of heart rate decrease will be than compared between patients with sympathetic and parasympathetic predominance measured prior to drug injection.

ELIGIBILITY:
Inclusion Criteria:

* patients assessed with American Society of Anesthesiologists' Physical Status Classification System as 1-2 status
* planned surgery under general anaesthesia

Exclusion Criteria:

* known sensitivity to remifentanil
* anticipated problems with tracheal intubation
* increased risk of aspiration
* diabetic patients
* patients taking medications with known influence on autonomic nervous system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-05; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Vagomimetic effect of RMFNT in reference to autonomic nervous system activity | before and after drug injection

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Wujtewicz, Principal Investigator — Department of Ophthalmology, Medical University of Gdańsk
Locations (1):
- Medical University of Gdansk, Gdansk, Poland